CLINICAL TRIAL: NCT01468129
Title: A Prospective, Randomized Controlled Trial to Evaluate the Efficacy of Cell Saver to Redue Blood Loss in One-stage Bilateral Total Hip Arthroplasty (THA)
Brief Title: Cell Saver Use in Bilateral Total Hip Arthroplasty (THA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Other Study IDs: 11UJPAR
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: One-stage Bilateral Total Hip Replacement
MeSH Terms: interventions — Operative Blood Salvage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cell Saver (Active Comparator)
  Interventions: Other: Cell Saver
- Non Cell Saver (No Intervention)

INTERVENTIONS:
Other: Cell Saver
  Arms: Cell Saver

SUMMARY:
This study will investigate the efficacy of using cell saver during bilater total hip arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Subject is over 21 years of age
* Subject with bilateral degenerative disease of hips who are candidate for one-stage bilateral THA
* Subject willing and able to provide written informed consent

Exclusion Criteria:

* Subject with significant comorbidities identified by Charleston index of ≥ 3
* Subject with malignancy
* Subject with history of heart disease, myocardial infarction, pulmonary insufficiency, pulmonary embolus, documented fat emboli syndrome, adult respiratory distress syndrome, documented patent ductus arteriosus or septal defect, chronic renal failure and/or acute hepatic failure or chirhosis
* Subjects with hematologic disorders such as anemia (Hb < 10 g/dL) and sickle cell disease, acquired or congenital coagulopathies, acquired or congenital bleeding disorders,
* Subject who received anticoagulant such as aspirin or Warfarin (Coumadin) or antiplatelet agents such as clopidogrel (Plavix) within 7 days of surgery
* Subject who received hemostatic agents such as tranexamic acid and aprotinin
* Subjects utilizing acute normovolumic haemodilution
* Subject is not permitted to remain without his/her anti-coagulant regimen (eg Plavix) for 48 hours postoperatively
* Subject is known to be pregnant.
* Subject has erythropoietin agonist/stimulating agent within 90 days prior to surgery.
* Presence of contaminants such as urine, fat, bowel contents, and most importantly infection in the operative field
* Presence of vasoactive drugs such as papaverine in the operative field

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-11; Primary Completion 2012-12; Study Completion 2012-12

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States